CLINICAL TRIAL: NCT04379167
Title: A Phase 2, Single Arm, Open Label Clinical Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of YY-20394 in Patients With Relapsed/Refractory Follicular Non-Hodgkin's Lymphoma Who Have Failed at Least Two Prior Systemic Therapies.
Brief Title: A Phase 2 Clinical Study of YY-20394 in Patients With Relapsed/Refractory Follicular Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-009
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 is a selective inhibitor of the delta isoform of phosphatidylinositol 3 kinase (PI3K-δ) which differs structurally from idelalisib, a PI3K-δ inhibitor approved for patients with relapsed chronic lymphocytic leukemia and indolent lymphoma.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — YY-20394 is a selective inhibitor of the delta isoform of phosphatidylinositol 3 kinase (PI3K-δ) which differs structurally from idelalisib, a PI3K-δ inhibitor approved for patients with relapsed chronic lymphocytic leukemia and indolent lymphoma. PI3K-δ signaling pathways are frequently hyperactive in B-cell cancers, making inhibition of PI3K-δ a promising target for B-cell malignancies. YY 20394 has high potency against PI3K-δ, but with markedly improved selectivity in in vitro assays compared to idelalisib. This higher selectivity for PI3K-δ may decrease the risk of serious infection seen with idelalisib and duvelisib (a PI3K-γ/δ dual inhibitor) due to strong immune suppression.

SUMMARY:
A Phase 2, single arm, open label clinical study to evaluate the efficacy, safety, tolerability and pharmacokinetics of YY-20394 as monotherapy in patients with relapsed/refractory follicular non-Hodgkin's lymphoma who have failed at least two prior systemic therapies

ELIGIBILITY:
Inclusion Criteria:

- Age

1. Patient is ≥18 years of age at the time of signing the informed consent. Type of Patient and Disease Characteristics
2. Has histologically confirmed follicular non-Hodgkin's lymphoma Grade ≤3 according to the WHO 2017 classification system.
3. Has radiographically measurable disease as per Lugano Criteria with at least one nodal lesion (which has not been previous radiated) that is >15 mm in long axis, regardless of the length of the short axis, AND/OR extranodal lesion of >10 mm in long and short axis.
4. Has received at least two prior lines of systemic therapy (excluding radiation) for follicular lymphoma. Refractory disease is defined as persistence of evaluable disease after therapy with documented disease progression at the time of enrollment.
5. Must have relapsed (experienced disease progression) during their last follicular lymphoma regimen after receiving at least two cycles of therapy or within 12 months after completing their last regimen for follicular lymphoma.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Has a life expectancy >3 months.
8. Has adequate organ function as defined in Table 5 1. Specimen for this assessment must be collected within 14 days prior to the first dose of study treatment:
9. Patient is male or female.
10. Male patients are eligible to participate if they agree to use a highly effective contraception as detailed in Appendix 4 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
11. Female patient are eligible to participate if they are not pregnant (see Appendix 4), not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4. OR
    * A WOCBP who agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent from heterosexual intercourse as their preferred method and usual lifestyle as described in Appendix 4, beginning 28 days before the start of study treatment, during the treatment period and for at least 3 months after the last dose of study treatment.
    * A WOCBP must have a negative serum pregnancy within 72 hours of the first dose of study treatment.
12. Patient is capable of giving signed informed consent as described in Appendix 1 (Section 10.1.3) which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
13. Must be willing and able to adhere to the study and lifestyle restrictions.

Exclusion Criteria:

1. Has follicular lymphoma histological Grade >3 or histologic evidence of transformation to a high-grade or diffuse large B-cell lymphoma.
2. Has presence of central nervous system (CNS) disease (either CNS lymphoma or leptomeningeal lymphoma) that is clinically uncontrolled or diagnosed within 4 months of enrollment.
3. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication.

   Note: During the treatment period, patients should not take medication that may prolong the QT (such as antiarrhythmic drugs).
4. Has peripheral neuropathy that is ≥Grade 2 with pain.
5. Has a medical history of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the study treatment.
6. Has diarrhea of CTCAE Grade >1.
7. Has a history of or concurrent interstitial lung disease of any severity and/or severely impaired lung function.
8. Prior history of drug-induced colitis or drug-induced pneumonitis.
9. Has a systemic infection or other serious infection requiring systemic treatment within 14 days before the first dose of study treatment.
10. Has a known additional malignancy that is progressing or required active treatment within 2 years of enrollment.

    Note: patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast, cervical cancer in situ, superficial bladder tumors [Ta and Tis; carcinoma in situ]) who have undergone curative therapy with no evidence of recurrence are not excluded.

    Prior/Concomitant Therapy
11. Has received prior treatment with YY-20394, or other PIK3-δ inhibitors.
12. Has received prior treatment with rituximab or other unconjugated antibody treatment within 28 days (21 days if clear evidence of progressive disease or immediate treatment is mandated) prior to the first dose of study treatment.
13. Has received radioimmunoconjugates or toxin conjugates within 12 weeks before the first dose of study treatment.
14. Has had received prior systemic anticancer therapy, or targeted small molecule therapy, or definitive radiotherapy ≤28 days (14 days for palliative radiation) prior to the first dose of study treatment.

    Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 alopecia may be eligible.

    Note: Patients must have recovered from all radiation-related toxicities.
15. Has undergone major surgery (excluding lymph node biopsy) or significant trauma ≤4 weeks before the first dose of study treatment.

    Note: patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study treatment.
16. Has had autologous stem cell transplant within 6 months prior to first dose of study treatment, or prior allograft stem cell transplantation at any time.
17. Use of medications or foods that are moderate cytochrome P (CYP)3A inhibitors, strong or moderate CYP3A inducers within 14 days prior to first dose of study treatment or 5 half-lives of the given drug, whichever is longer.
18. Has a history of immunodeficiency or has received systemic steroids (in dosing exceeding 10 mg daily of prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days of the first dose of study treatment. The use of physiological doses of corticosteroids may be approved after consultation with the Sponsor.
19. Has received a live vaccination within 4 weeks before the first dose of study treatment. Examples of live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster, yellow fever, Bacille Calmette-Guérin (BCG) and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
20. Has received granulocyte colony-stimulating factor or blood transfusion within 7 days before start of screening.

    Prior/Concurrent Clinical Study Experience
21. Is currently participating in or has participated in a study with an investigational compound or device within ≤4 weeks prior to the first dose of study treatment.

    Note: Patients who have entered the follow-up phase of an investigational study may participate so long as it has been at least 4 weeks since the last dose of the previous investigational agent.

    Diagnostic Assessments
22. Has a known history of or newly diagnosed infection with HIV, Hepatitis B (defined as HBsAg reactive) or hepatitis C virus (HCV) (defined as detection of qualitative HCV virus RNA).
23. Has a history or current evidence of any condition, laboratory abnormality or other circumstances that might confound the results of the study or interfere with participation for the full duration of the study, such that it is not in the best interests of the patient to take part in the study.

    Other Exclusions
24. Patient is pregnant or breastfeeding or expecting to conceive of father children for the duration of the study.
25. Has a history of hypersensitivity to YY-20394 and/or any excipients.
26. Has a history of hypersensitivity to radiological imaging contrasting agents.
27. Has a known psychiatric disorder that would interfere with proper cooperation with the requirements of the study.
28. Is a regular user of illicit or recreational drugs or has had a recent history (within the last year) of drug or alcohol abuse of dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) | throughout the study approximately 2 years
  complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
evaluate duration of response (DOR) | throughout the study approximately 2 years
  DOR, defined as time from first documentation of a response (PR or CR) to the first documented disease progression or death due to any cause, whichever occurs first, for those patients with a PR or CR.

OTHER OUTCOMES:
progression-free survival (PFS) | throughout the study approximately 2 years
  the time from the first dose of study treatment to first documented disease progression or death due to any cause, whichever occurs first.
Adverse events (AEs) | throughout the study approximately 2 years
  Adverse events refer to all adverse medical events occurred after the subject received the test drug
AUClast | throughout the study approximately 2 years
  • Area under the plasma concentration-time curve from time zero to time of last measurable concentration
AUCinf | throughout the study approximately 2 years
  • Area under the plasma concentration-time curve from time zero extrapolated to infinite time
Cmin | throughout the study approximately 2 years
  Minimum observed concentration
Cmax | throughout the study approximately 2 years
  Maximum observed concentration
Half-life (T1/2) | throughout the study approximately 2 years
  The time it takes to reduce the concentration of drugs in the blood or the amount of drugs in the body to one-half
Time to Cmax (Tmax) | tThe time when the blood concentration reaches the peak value after a single administration.hroughout the study approximately 2 years

IPD SHARING:
Plan to Share IPD: Yes
The plan to make individual participant data (IPD) available to still remains uncertain.
Supporting Information: CSR
Time Frame: After the clinical trail.
Access Criteria: It will be updated later.